CLINICAL TRIAL: NCT01636206
Title: A Phase 3, Multicenter, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Safety of a 5.0% Concentration of Lifitegrast Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye (SONATA)
Brief Title: Safety Study of Lifitegrast to Treat Dry Eye
Acronym: SONATA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1118-DRY-400
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Lifitegrast (Experimental): Active
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — Dosage Form: Ophthalmic Solution Dosage: 5.0% Frequency: BID Duration: ~1 year
  Arms: Lifitegrast
Drug: Placebo — Dosage Form: Ophthalmic Solution Dosage: placebo Frequency: BID Duration: ~1 year
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety of lifitegrast ophthalmic solution compared to placebo in the treatment of dry eye as assessed by ocular and non-ocular adverse events when administered BID for approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, sign and date the informed consent and HIPAA documents
* Willing and able to comply with all study procedures
* Be at least 18 years of age
* Patient-reported history of dry eye in both eyes
* A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period

Exclusion Criteria:

* Any ocular condition that, in the opinion of the Investigator, could affect study parameters including, but not limited to, active ocular infection, ocular inflammation, glaucoma, and/or diabetic retinopathy
* Unwilling to avoid wearing contact lenses for 24h prior to Visit 1 and for some duration during the study
* Any blood donation or significant loss of blood within 56 days of Visit 1
* Any history of immunodeficiency disorder, positive HIV, hepatitis B, C, or evidence of acute active hepatitis A (anti-HAV IgM), or organ or bone marrow transplant.
* Use of any prohibited medications during the appropriate pre-study washout period and at any time during the study unless otherwise specified
* Any significant illness that could interfere with study parameters
* History of laser-assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery within 12 months prior to Visit 1, and/or any other ocular surgical procedure within 12 months prior to Visit 1; or any scheduled ocular surgical procedure during the study period.
* Known history of alcohol and/or drug abuse
* Subjects with Dry eye secondary to scarring or destruction of conjunctival goblet cells (as with Vitamin A deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2014-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (23):
  - SONATA Investigational Site, Artesia, California
  - SONATA Investigational Site, Hemet, California
  - SONATA Investigational Site, Laguna Hills, California
  - SONATA Investigational Site, Lancaster, California
  - SONATA Investigational Site, Montebello, California
  - SONATA Investigational Site, Parker, Colorado
  - SONATA Investigational Site, Boynton Beach, Florida
  - SONATA Investigational Site, Roswell, Georgia
  - SONATA Investigational Site, Hoffman Estates, Illinois
  - SONATA Investigational Site, Edgewood, Kentucky
  - SONATA Investigational Site, Lexington, Kentucky
  - SONATA Investigational Site, Stillwater, Minnesota
  - SONATA Investigational Site, Pennington, New Jersey
  - SONATA Investigational Site, Woodland Park, New Jersey
  - SONATA Investigational Site, Rochester, New York
  - SONATA Investigational Site, Rockville Centre, New York
  - SONATA Investigational Site, Charlotte, North Carolina
  - SONATA Investigational Site, High Point, North Carolina
  - SONATA Investigational Site, Cleveland, Ohio
  - SONATA Investigational Site, Doylestown, Pennsylvania
  - SONATA Investigational Site, Mt. Pleasant, South Carolina
  - SONATA Investigational Site, Chattanooga, Tennessee
  - SONATA Investigational Site, Houston, Texas

REFERENCES:
- [Result] Donnenfeld ED, Karpecki PM, Majmudar PA, Nichols KK, Raychaudhuri A, Roy M, Semba CP. Safety of Lifitegrast Ophthalmic Solution 5.0% in Patients With Dry Eye Disease: A 1-Year, Multicenter, Randomized, Placebo-Controlled Study. Cornea. 2016 Jun;35(6):741-8. doi: 10.1097/ICO.0000000000000803. PMID 27055211

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Lifitegrast
Started | 111 | 221
Completed | 92 | 170
Not Completed | 19 | 51

BASELINE CHARACTERISTICS:
Population: Randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lifitegrast | Total
Number analyzed (Participants) | 111 | 221 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (13.18) | 58.8 (12.39) | 59.5 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 165 | 250
  Male | 26 | 56 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular and Nonocular Treatment Emergent Adverse Events (TEAEs) for 1 Year
Time Frame: Day 0 to Day 360
Population: Safety population included all randomized participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Lifitegrast
Number analyzed (Participants) | 111 | 220
participants
  Ocular TEAE | 38 | 118
  Non-ocular TEAE | 40 | 104

ADVERSE EVENTS:
Arm/Group | Placebo | Lifitegrast
Serious Adverse Events (participants affected / at risk) | 6/111 | 9/220
Other Adverse Events (participants affected / at risk) | 22/111 | 92/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | Lifitegrast (N=220)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colonic polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | Lifitegrast (N=220)
Dry eye (Eye disorders) | 6 (6) | 4 (4)
Visual acuity reduced (Eye disorders) | 7 (8) | 25 (28)
Instillation site irritation (General disorders) | 5 (5) | 33 (33)
Instillation site reaction (General disorders) | 2 (2) | 29 (30)
Dysgeusia (Nervous system disorders) | 2 (2) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.